CLINICAL TRIAL: NCT02384265
Title: Financial Incentives and SMS to Improve African American Womens' Glycemic Control: Friends & Relatives Improving the Effectiveness of Networks for Diabetes Support Through Text Messaging (FRIENDS Text)
Brief Title: Financial Incentives and Text Messaging to Improve African American Womens' Glycemic Control
Acronym: FRIENDS-Text
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Arleen F. Brown, MD, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1P60MD006923 (NIH)
Record Dates: First submitted 2015-02-25; First posted 2015-03-10 (Estimated); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Disparities; Behavioral; Text messaging; Social networks; African American; Female
MeSH Terms: conditions — Diabetes Mellitus; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IM/SMS + Incentive Condition (Experimental): Participants in the intervention condition will consist of the PWD and their two STMs. The PWD and STM will receive the same protocols that the "Usual Care" participants receive, including an introductory educational session, written materials on diabetes, a blood glucose log, and a physical activity monitoring log. The PWDs in this condition will also receive training in action planning with their STMs. They will also receive SMS messages supporting diabetes self-care from the study team. The study team will also encourage the STMs to interaction in person and via text messages with the PWD.
  Interventions: Behavioral: IM/SMS + Incentive Condition
- Control (No Intervention): Control group participants will consist of the person with diabetes (PWD) and their two support team members (STM). The PWD will receive regular medical care from their usual providers. They will also receive an introductory educational session and written materials on diabetes, the importance of its control, and diabetes self-care strategies, and a blood glucose and physical activity monitoring log. They will be invited for study visits at 3, 6, and 12 months to measure cholesterol, A1c (for those with diabetes), blood pressure, height, and weight measurement. PWDs and STMs in the control condition will receive generic health promotion information during in-person visits or by mail. They will receive follow-up messages by text to remind them about study related events.

INTERVENTIONS:
Behavioral: IM/SMS + Incentive Condition — See description of Intervention arm protocols above.
  Arms: IM/SMS + Incentive Condition

SUMMARY:
Diabetes is a major public health problem that is associated with substantial health disparities for African American women compared to African American men or white men and women. This project will incorporate a) new technology whose use is high among African Americans (cell phone text message reminders), b) support from social networks, and c) strategies from the emerging field of behavioral economics to encourage and support self care behaviors that lead to improvements in diabetes control.

In Stage I of the study, the investigators conducted focus groups with women with diabetes and their family members and friends. The investigators used information from these groups to work with a team of community partners to develop recruitment protocols, prepare study documents (including flyers, Frequently Asked Questions sheets, and informed consent forms), and finalize participant surveys.

In the next phase of the study the investigators will evaluate ways that friends and family members can use direct support and text messages to improve control of blood sugar for African American women with type 2 diabetes. A team of three people--the Person With Diabetes (PWD) and 2 friends or family members, also known as the Support Team Members (STMs)--will be assigned at random to one of two groups to compare approaches to improving control of blood sugar. Each team will receive information and resources on improving diabetes control and will be linked by a text messaging program. The intervention team will receive additional text messaging support that may help them improve the PWD's diabetes control.

DETAILED DESCRIPTION:
Control Condition. Control group participants will consist of the person with diabetes (PWD) and their two support team members (STMs). The PWD will receive regular medical care from their usual providers. They will also receive an introductory educational session and written materials on diabetes, the importance of its control, and diabetes self-care strategies, and a blood glucose and physical activity monitoring log. They will be invited for study visits, distinct from their routine clinic visits, at 3, 6, and 12 months to measure cholesterol, A1c (for those with diabetes), blood pressure, height, and weight measurement. Participants in the control condition will receive generic health promotion information during in-person visits or by mail. They will receive follow-up messages by text to remind them about study related events.

Intervention Group. Participants in the intervention condition will consist of the PWD and their two STMs. The PWD will receive the same protocols that the "Usual Care" participants receive, including an introductory educational session, written materials on diabetes, a blood glucose log, and a physical activity monitoring log.

The PWDs in the intervention group will receive training in action planning that is linked to their role self-identity. Role identity will be kept highly salient throughout the study by using identity primes that remind the individual that both processes (diabetes self-care behaviors) and goals (achieving A1c targets) are important responsibilities associated with that role. For example, participants may be asked to keep a picture or memento that reminds them of their role identity (e.g., a picture of a child or a photo of a place she would like to visit) on a blood sugar and physical activity log that the study will provide to the patient. The STMs in the intervention group will discuss these role identities and motivators with the PWD in their team intake session. They will also obtain similar training in action planning and in ways to support the PWD in order to better control her diabetes.

Intervention team members will be reminded of the PWD's intrinsic motivations (IM), and how engaging in regular diabetes self-care can improve diabetes control, during interactions designed to boost the participants' confidence that they can accomplish and sustain the behavior change that contributes to interim and longer term goals. These interactions include text messages between the support team and the study team and between members of the support team. The text messages will include individually- and/or culturally-tailored messages, some of which are linked to the motivating factors identified through the questionnaire and probes. The text messages will take varying forms: (a) General diabetes messages derived from sources such as the ADA African American Programs and the National Diabetes Education Program; (b) Reminders about blood glucose monitoring, medication adherence, diet, and exercise, and how these behaviors contribute to maintaining role identity; (c) Prompts or queries about home glucose monitor readings and their frequencies that allow participants to communicate by text with study staff on non-urgent matters; and (d) Challenges and contests for which they receive supportive text messages.

Face-to-Face Meetings will occur at the baseline and months 3, 6, and 12 to gather study data. For the intervention group, this will also include contact with a study team member who helps the intervention PWD and STMs identify and agree to desired behaviors and A1c targets. The study team member will review glucometer readings, medication refills, and A1c levels; encourage each PWD to engage in processes (e.g., self-monitoring or adhering to medications); encourage STMs in their supportive roles; congratulate those PWDs who near or reach A1c targets; and motivate those having difficulty reaching their targets.

Baseline Protocols and Data Collection After randomization, all participants will be asked to provide verbal consent for the survey tailored to their study arm and their role as a PWD or STM, and will be administered a 35-45 minute baseline in-person survey in English by phone. There will be four different versions of the survey: Intervention PWD, Intervention STM, Control PWD, and Control STM. Following the administration of the baseline survey, all intervention participants will be allowed to select the message themes that they would like to receive from a list of options based on factors that they identified as intrinsic motivators and the intervals at which they would like to receive text messages (range 5 per week to 2 per day). The investigators plan to send an average of three messages per day, and elicit on average 1-2 responses per day. Additionally, the intervention PWDs will be told their target A1c goals and the incentives associated with specific drops in A1c. At this stage, the study staff will again discuss with the PWDs and STMs intervention groups the potential risks and harms of using inappropriate strategies to try to attain glycemic targets and, to obtain the monetary incentives. All enrolled patients will participate in a small group 30 minute session with study staff in the clinic to discuss diabetes self-care. All participants will also be invited to participate in ongoing diabetes classes and activities, and each person will be given a list of diabetes resources available in their clinic (e.g. group and individual diabetes education) and a calendar of local events and activities, such as the ADA Project Power diabetes classes in local churches, exercise classes, and healthy eating groups.

Follow-up Protocols and Data Collection Once a month for the 6 month intervention period, participants in the intervention groups will receive a phone call from study staff to reinforce intrinsic motivation for improved glycemic control. At months 3, 6, and 12, participants (PWDs) in the control and intervention group will receive a reminder that the A1c test is due (via phone, mail, and text message). At months 3 and 6, the intervention team will also receive a message (via phone, mail, and text) about the deadline for an in-person incentive payment. In addition, intervention participants (PWDs) who attain target A1c levels will receive the appropriate monetary incentives based on their new A1c levels and through participation in the lottery. Compensation and incentives will be delivered at the time of testing. At the 6 month visit, all study subjects in both groups will be administered an abbreviated version of the baseline survey. At this point the financial incentives will be withdrawn and the IM, reminder, and generic text messages will stop for the intervention arm, who, like the control arm, will only receive reminder messages for clinic visits to get A1c tested (A1c testing will only be completed with PWDs in the control and intervention groups). At 12 months, all PWD and STM participants will complete a final survey. In the event the investigators are unable to reach the study participants, the investigators will obtain alternate contact information during study enrollment for all participants using a locator form. This form will be stored separate from the study participants' data. This will help to increase retention over the course of the study, and the investigators will update contact information regularly via the text messages. Once the 12-month study visit has been completed, the locator form will be destroyed.

Assess the costs of the interventions In order to determine feasibility of importing the results of this study into public community clinics a costs analysis is planned at the end of the study. Costs fall into two main categories: program costs and costs of health services used by study participants. Program costs will be based on actual costs incurred by the study, including staff time and supplies, as well as the opportunity cost of time incurred by participants for attending quarterly study visits and participating in study phone calls. Costs related to personnel time will be measured as the product of personnel time spent and unit cost of labor and fringe benefits for the study staff. Personnel time spent for each study condition will be estimated from self-report. Costs related to use of resources (equipment and supplies, overhead) will be measured as the product of quantities used and unit cost derived from accounting data. The program developmental and training costs will be measured, but will be divided equally for the two intervention arms since identical protocols and provider trainings are required in each arm. Costs that are solely for research purpose, such as data management and analysis, will be excluded. The investigators will derive health services costs from survey data collected in the surveys from all study participants. These data include information on the number of outpatient medical visits, hospital stays, and Emergency Department visits. Using data in the published literature (e.g. using Medicare data), the investigators will map costs onto units of utilization, such as the cost for one physician office visit or one day in the hospital, thereby allowing the investigators to estimate total costs incurred for health services.

ELIGIBILITY:
Inclusion Criteria:

* Eligible persons with diabetes (PWDs) will be identified either through the clinic diabetes registry, referrals from their providers, or direct recruitment by study staff during clinic hours. Eligible subjects are African American women seen at the clinic at least once in the prior 12 months, who have a record of at least one A1c reading in the past year (most recent A1c >8%), indicate that they plan to receive their diabetes care from the clinic over the next 18 months, and have a cell phone with an active plan, have two other individuals who they identify as friends or family members to enroll with them.
* Eligible support team members (STMs) will be identified by the PWD as being a friend or family member 18 years or older and have a cell phone with an active plan.
* To enroll in the study, there must be a triad (1 PWD and 2 STMs) that meet all study inclusion requirements. After the study begins, if one of the STMs drops out/withdrawals from the study, the team can continue to participate. However, if the PWD drops out/withdrawals from the study, the team will not be able to continue in the study and therefore, will be dropped from the study by the principal investigator.

Exclusion Criteria:

* The investigators will exclude PWDs who are pregnant at the time of enrollment or those who only had diabetes during pregnancy, children, prisoners, homeless persons, institutionalized adults, and adults with type 1 diabetes, hemophilia, AIDS, cancer, hemoglobinopathies, or severe mental illness.
* The investigators will exclude STMs who are younger than 18 years old or do not have a cell phone with an active plan.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06-21; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c at 12-months | 12-months
  The investigators will measure the change in hemoglobin A1c (measured as % A1c).

SECONDARY OUTCOMES:
Change from Baseline in Weight 12-months | 12 months
  The investigators will measure the change in weight (measured in kg).
Change from Baseline in Body Mass Index at 12-months | 12 months
  The investigators will measure the change in Body Mass Index (measured in kg/meter2).
Change from Baseline in Waist Circumference (inches) at 12-months | 12 months
  The investigators will measure the change in waist circumference (measured in centimeters).
Change from Baseline in Systolic and Diastolic Blood Pressure at 12-months | 12 months
  The investigators will measure the change in systolic and diastolic blood pressure measured in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Arleen F Brown, M.D., Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Holman United Methodist Church, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacks DB, Bruns DE, Goldstein DE, Maclaren NK, McDonald JM, Parrott M. Guidelines and recommendations for laboratory analysis in the diagnosis and management of diabetes mellitus. Clin Chem. 2002 Mar;48(3):436-72. PMID 11861436
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Ohkubo Y, Kishikawa H, Araki E, Miyata T, Isami S, Motoyoshi S, Kojima Y, Furuyoshi N, Shichiri M. Intensive insulin therapy prevents the progression of diabetic microvascular complications in Japanese patients with non-insulin-dependent diabetes mellitus: a randomized prospective 6-year study. Diabetes Res Clin Pract. 1995 May;28(2):103-17. doi: 10.1016/0168-8227(95)01064-k. PMID 7587918
- [Background] Grant R, Adams AS, Trinacty CM, Zhang F, Kleinman K, Soumerai SB, Meigs JB, Ross-Degnan D. Relationship between patient medication adherence and subsequent clinical inertia in type 2 diabetes glycemic management. Diabetes Care. 2007 Apr;30(4):807-12. doi: 10.2337/dc06-2170. Epub 2007 Jan 26. PMID 17259469
- [Background] Grant RW, Cagliero E, Dubey AK, Gildesgame C, Chueh HC, Barry MJ, Singer DE, Nathan DM, Meigs JB. Clinical inertia in the management of Type 2 diabetes metabolic risk factors. Diabet Med. 2004 Feb;21(2):150-5. doi: 10.1111/j.1464-5491.2004.01095.x. PMID 14984450
- [Background] Brown AF, Gregg EW, Stevens MR, Karter AJ, Weinberger M, Safford MM, Gary TL, Caputo DA, Waitzfelder B, Kim C, Beckles GL. Race, ethnicity, socioeconomic position, and quality of care for adults with diabetes enrolled in managed care: the Translating Research Into Action for Diabetes (TRIAD) study. Diabetes Care. 2005 Dec;28(12):2864-70. doi: 10.2337/diacare.28.12.2864. PMID 16306546
- [Background] Heisler M, Smith DM, Hayward RA, Krein SL, Kerr EA. Racial disparities in diabetes care processes, outcomes, and treatment intensity. Med Care. 2003 Nov;41(11):1221-32. doi: 10.1097/01.MLR.0000093421.64618.9C. PMID 14583685
- [Background] Harris MI, Eastman RC, Cowie CC, Flegal KM, Eberhardt MS. Racial and ethnic differences in glycemic control of adults with type 2 diabetes. Diabetes Care. 1999 Mar;22(3):403-8. doi: 10.2337/diacare.22.3.403. PMID 10097918
- [Background] Karter AJ, Ferrara A, Liu JY, Moffet HH, Ackerson LM, Selby JV. Ethnic disparities in diabetic complications in an insured population. JAMA. 2002 May 15;287(19):2519-27. doi: 10.1001/jama.287.19.2519. PMID 12020332
- [Background] Peek ME, Cargill A, Huang ES. Diabetes health disparities: a systematic review of health care interventions. Med Care Res Rev. 2007 Oct;64(5 Suppl):101S-56S. doi: 10.1177/1077558707305409. PMID 17881626
- [Background] Sequist TD, Fitzmaurice GM, Marshall R, Shaykevich S, Marston A, Safran DG, Ayanian JZ. Cultural competency training and performance reports to improve diabetes care for black patients: a cluster randomized, controlled trial. Ann Intern Med. 2010 Jan 5;152(1):40-6. doi: 10.7326/0003-4819-152-1-201001050-00009. PMID 20048271
- [Background] Lussier JP, Heil SH, Mongeon JA, Badger GJ, Higgins ST. A meta-analysis of voucher-based reinforcement therapy for substance use disorders. Addiction. 2006 Feb;101(2):192-203. doi: 10.1111/j.1360-0443.2006.01311.x. PMID 16445548
- [Background] Malotte CK, Rhodes F, Mais KE. Tuberculosis screening and compliance with return for skin test reading among active drug users. Am J Public Health. 1998 May;88(5):792-6. doi: 10.2105/ajph.88.5.792. PMID 9585747
- [Background] Seal KH, Kral AH, Lorvick J, McNees A, Gee L, Edlin BR. A randomized controlled trial of monetary incentives vs. outreach to enhance adherence to the hepatitis B vaccine series among injection drug users. Drug Alcohol Depend. 2003 Aug 20;71(2):127-31. doi: 10.1016/s0376-8716(03)00074-7. PMID 12927650
- [Background] Stevens-Simon C, O'Connor P, Bassford K. Incentives enhance postpartum compliance among adolescent prenatal patients. J Adolesc Health. 1994 Jul;15(5):396-9. doi: 10.1016/1054-139x(94)90263-1. PMID 7947854
- [Background] Donatelle R, Hudson D, Dobie S, Goodall A, Hunsberger M, Oswald K. Incentives in smoking cessation: status of the field and implications for research and practice with pregnant smokers. Nicotine Tob Res. 2004 Apr;6 Suppl 2:S163-79. doi: 10.1080/14622200410001669196. PMID 15203819
- [Background] Hey K, Perera R. Competitions and incentives for smoking cessation. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD004307. doi: 10.1002/14651858.CD004307.pub2. PMID 15846705
- [Background] Volpp KG, Troxel AB, Pauly MV, Glick HA, Puig A, Asch DA, Galvin R, Zhu J, Wan F, DeGuzman J, Corbett E, Weiner J, Audrain-McGovern J. A randomized, controlled trial of financial incentives for smoking cessation. N Engl J Med. 2009 Feb 12;360(7):699-709. doi: 10.1056/NEJMsa0806819. PMID 19213683
- [Background] Volpp KG, Loewenstein G, Troxel AB, Doshi J, Price M, Laskin M, Kimmel SE. A test of financial incentives to improve warfarin adherence. BMC Health Serv Res. 2008 Dec 23;8:272. doi: 10.1186/1472-6963-8-272. PMID 19102784
- [Background] Volpp KG, John LK, Troxel AB, Norton L, Fassbender J, Loewenstein G. Financial incentive-based approaches for weight loss: a randomized trial. JAMA. 2008 Dec 10;300(22):2631-7. doi: 10.1001/jama.2008.804. PMID 19066383
- [Background] Curry SJ, Wagner EH, Grothaus LC. Evaluation of intrinsic and extrinsic motivation interventions with a self-help smoking cessation program. J Consult Clin Psychol. 1991 Apr;59(2):318-24. doi: 10.1037//0022-006x.59.2.318. PMID 2030194
- [Background] Williams GC, Gagne M, Ryan RM, Deci EL. Facilitating autonomous motivation for smoking cessation. Health Psychol. 2002 Jan;21(1):40-50. PMID 11846344
- [Background] Williams GC, McGregor HA, Zeldman A, Freedman ZR, Deci EL. Testing a self-determination theory process model for promoting glycemic control through diabetes self-management. Health Psychol. 2004 Jan;23(1):58-66. doi: 10.1037/0278-6133.23.1.58. PMID 14756604
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Cowie CC, Rust KF, Ford ES, Eberhardt MS, Byrd-Holt DD, Li C, Williams DE, Gregg EW, Bainbridge KE, Saydah SH, Geiss LS. Full accounting of diabetes and pre-diabetes in the U.S. population in 1988-1994 and 2005-2006. Diabetes Care. 2009 Feb;32(2):287-94. doi: 10.2337/dc08-1296. Epub 2008 Nov 18. PMID 19017771
- [Background] Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications Research Group; Lachin JM, Genuth S, Cleary P, Davis MD, Nathan DM. Retinopathy and nephropathy in patients with type 1 diabetes four years after a trial of intensive therapy. N Engl J Med. 2000 Feb 10;342(6):381-9. doi: 10.1056/NEJM200002103420603. PMID 10666428
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Brown AF, Gerzoff RB, Karter AJ, Gregg E, Safford M, Waitzfelder B, Beckles GL, Brusuelas R, Mangione CM; TRIAD Study Group. Health behaviors and quality of care among Latinos with diabetes in managed care. Am J Public Health. 2003 Oct;93(10):1694-8. doi: 10.2105/ajph.93.10.1694. PMID 14534224
- [Background] Heisler M, Faul JD, Hayward RA, Langa KM, Blaum C, Weir D. Mechanisms for racial and ethnic disparities in glycemic control in middle-aged and older Americans in the health and retirement study. Arch Intern Med. 2007 Sep 24;167(17):1853-60. doi: 10.1001/archinte.167.17.1853. PMID 17893306
- [Background] Duru OK, Gerzoff RB, Selby JV, Brown AF, Ackermann RT, Karter AJ, Ross S, Steers N, Herman WH, Waitzfelder B, Mangione CM. Identifying risk factors for racial disparities in diabetes outcomes: the translating research into action for diabetes study. Med Care. 2009 Jun;47(6):700-6. doi: 10.1097/mlr.0b013e318192609d. PMID 19480090
- [Background] Hofer TP, Hayward RA, Greenfield S, Wagner EH, Kaplan SH, Manning WG. The unreliability of individual physician "report cards" for assessing the costs and quality of care of a chronic disease. JAMA. 1999 Jun 9;281(22):2098-105. doi: 10.1001/jama.281.22.2098. PMID 10367820
- [Background] Krein SL, Hofer TP, Kerr EA, Hayward RA. Whom should we profile? Examining diabetes care practice variation among primary care providers, provider groups, and health care facilities. Health Serv Res. 2002 Oct;37(5):1159-80. doi: 10.1111/1475-6773.01102. PMID 12479491
- [Background] Piette JD, Heisler M, Harand A, Juip M. Beliefs about prescription medications among patients with diabetes: variation across racial groups and influences on cost-related medication underuse. J Health Care Poor Underserved. 2010 Feb;21(1):349-61. doi: 10.1353/hpu.0.0247. PMID 20173274
- [Background] Coleman K, Reiter KL, Fulwiler D. The impact of pay-for-performance on diabetes care in a large network of community health centers. J Health Care Poor Underserved. 2007 Nov;18(4):966-83. doi: 10.1353/hpu.2007.0090. PMID 17982218
- [Background] Millett C, Gray J, Bottle A, Majeed A. Ethnic disparities in blood pressure management in patients with hypertension after the introduction of pay for performance. Ann Fam Med. 2008 Nov-Dec;6(6):490-6. doi: 10.1370/afm.907. PMID 19001300
- [Background] Millett C, Gray J, Saxena S, Netuveli G, Khunti K, Majeed A. Ethnic disparities in diabetes management and pay-for-performance in the UK: the Wandsworth Prospective Diabetes Study. PLoS Med. 2007 Jun;4(6):e191. doi: 10.1371/journal.pmed.0040191. PMID 17564486
- [Background] Millett C, Netuveli G, Saxena S, Majeed A. Impact of pay for performance on ethnic disparities in intermediate outcomes for diabetes: a longitudinal study. Diabetes Care. 2009 Mar;32(3):404-9. doi: 10.2337/dc08-0912. Epub 2008 Dec 10. PMID 19073759
- [Background] Deci EL, Koestner R, Ryan RM. A meta-analytic review of experiments examining the effects of extrinsic rewards on intrinsic motivation. Psychol Bull. 1999 Nov;125(6):627-68; discussion 692-700. doi: 10.1037/0033-2909.125.6.627. PMID 10589297
- [Background] Deci EL, Ryan RM. Intrinsic Motivation and Self-Determination in Human Behavior (Perspectives in Social Psychology). New York: Plenum Press; 1985.
- [Background] Greene D, Lepper MR. Effects of extrinsic rewards on children's subsequent intrinsic interest. Child Dev. 1974 Dec;45(4):1141-5. No abstract available. PMID 4143868
- [Background] Lorence D, Park H. Group disparities and health information: a study of online access for the underserved. Health Informatics J. 2008 Mar;14(1):29-38. doi: 10.1177/1460458207086332. PMID 18258673
- [Background] Lorence DP, Park H, Fox S. Racial disparities in health information access: resilience of the Digital Divide. J Med Syst. 2006 Aug;30(4):241-9. doi: 10.1007/s10916-005-9003-y. PMID 16978003
- [Background] Brown AF. Patient, system and clinician level interventions to address disparities in diabetes care. Curr Diabetes Rev. 2007 Nov;3(4):244-8. doi: 10.2174/157339907782329988. PMID 18220681
- [Background] Berger CC. Control of color of crowns for pulpless anterior teeth. J Prosthet Dent. 1968 Jan;19(1):58-9. doi: 10.1016/0022-3913(68)90010-3. No abstract available. PMID 5234948
- [Background] Duru OK, Mangione CM, Steers NW, Herman WH, Karter AJ, Kountz D, Marrero DG, Safford MM, Waitzfelder B, Gerzoff RB, Huh S, Brown AF; TRIAD Study Group. The association between clinical care strategies and the attenuation of racial/ethnic disparities in diabetes care: the Translating Research Into Action for Diabetes (TRIAD) Study. Med Care. 2006 Dec;44(12):1121-8. doi: 10.1097/01.mlr.0000237423.05294.c0. PMID 17122717
- [Background] Ettner SL, Cadwell BL, Russell LB, Brown A, Karter AJ, Safford M, Mangione C, Beckles G, Herman WH, Thompson TJ; TRIAD Study Group. Investing time in health: do socioeconomically disadvantaged patients spend more or less extra time on diabetes self-care? Health Econ. 2009 Jun;18(6):645-63. doi: 10.1002/hec.1394. PMID 18709636
- [Background] Gary TL, Safford MM, Gerzoff RB, Ettner SL, Karter AJ, Beckles GL, Brown AF. Perception of neighborhood problems, health behaviors, and diabetes outcomes among adults with diabetes in managed care: the Translating Research Into Action for Diabetes (TRIAD) study. Diabetes Care. 2008 Feb;31(2):273-8. doi: 10.2337/dc07-1111. Epub 2007 Nov 13. PMID 18000180
- [Background] Gregg EW, Karter AJ, Gerzoff RB, Safford M, Brown AF, Tseng CW, Waitzfielder B, Herman WH, Mangione CM, Selby JV, Thompson TJ, Dudley RA. Characteristics of insured patients with persistent gaps in diabetes care services: the Translating Research into Action for Diabetes (TRIAD) study. Med Care. 2010 Jan;48(1):31-7. doi: 10.1097/MLR.0b013e3181bd4783. PMID 20009778
- [Background] Karter AJ, Stevens MR, Brown AF, Duru OK, Gregg EW, Gary TL, Beckles GL, Tseng CW, Marrero DG, Waitzfelder B, Herman WH, Piette JD, Safford MM, Ettner SL. Educational disparities in health behaviors among patients with diabetes: the Translating Research Into Action for Diabetes (TRIAD) Study. BMC Public Health. 2007 Oct 29;7:308. doi: 10.1186/1471-2458-7-308. PMID 17967177
- [Background] Karter AJ, Stevens MR, Gregg EW, Brown AF, Tseng CW, Marrero DG, Duru OK, Gary TL, Piette JD, Waitzfelder B, Herman WH, Beckles GL, Safford MM, Ettner SL. Educational disparities in rates of smoking among diabetic adults: the translating research into action for diabetes study. Am J Public Health. 2008 Feb;98(2):365-70. doi: 10.2105/AJPH.2005.083501. Epub 2007 Jun 28. PMID 17600269
- [Background] Karter AJ, Stevens MR, Herman WH, Ettner S, Marrero DG, Safford MM, Engelgau MM, Curb JD, Brown AF; Translating Research Into Action for Diabetes Study Group. Out-of-pocket costs and diabetes preventive services: the Translating Research Into Action for Diabetes (TRIAD) study. Diabetes Care. 2003 Aug;26(8):2294-9. doi: 10.2337/diacare.26.8.2294. PMID 12882851
- [Background] Mangione CM, Gerzoff RB, Williamson DF, Steers WN, Kerr EA, Brown AF, Waitzfelder BE, Marrero DG, Dudley RA, Kim C, Herman W, Thompson TJ, Safford MM, Selby JV; TRIAD Study Group. The association between quality of care and the intensity of diabetes disease management programs. Ann Intern Med. 2006 Jul 18;145(2):107-16. doi: 10.7326/0003-4819-145-2-200607180-00008. PMID 16847293
- [Background] Selby JV, Swain BE, Gerzoff RB, Karter AJ, Waitzfelder BE, Brown AF, Ackermann RT, Duru OK, Ferrara A, Herman W, Marrero DG, Caputo D, Narayan KM; TRIAD Study Group. Understanding the gap between good processes of diabetes care and poor intermediate outcomes: Translating Research into Action for Diabetes (TRIAD). Med Care. 2007 Dec;45(12):1144-53. doi: 10.1097/MLR.0b013e3181468e79. PMID 18007164
- [Background] TRIAD Study Group. The Translating Research Into Action for Diabetes (TRIAD) study: a multicenter study of diabetes in managed care. Diabetes Care. 2002 Feb;25(2):386-9. doi: 10.2337/diacare.25.2.386. No abstract available. PMID 11815515
- [Background] Arsie MP, Marchioro L, Lapolla A, Giacchetto GF, Bordin MR, Rizzotti P, Fedele D. Evaluation of diagnostic reliability of DCA 2000 for rapid and simple monitoring of HbA1c. Acta Diabetol. 2000 Mar;37(1):1-7. doi: 10.1007/s005920070028. PMID 10928229
- [Background] Lenters-Westra E, Slingerland RJ. Six of eight hemoglobin A1c point-of-care instruments do not meet the general accepted analytical performance criteria. Clin Chem. 2010 Jan;56(1):44-52. doi: 10.1373/clinchem.2009.130641. Epub 2009 Nov 19. PMID 19926777
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Hackman J, Oldham G. Motivation through Design of Work-Test of a Theory. Organizational Behavior and Human Performance. 1976 1976;16:250-279.
- [Background] Heath C, Larrick RP, Wu G. Goals as reference points. Cogn Psychol. 1999 Feb;38(1):79-109. doi: 10.1006/cogp.1998.0708. PMID 10090799
- [Background] Krousel-Wood M, Islam T, Webber LS, Re RN, Morisky DE, Muntner P. New medication adherence scale versus pharmacy fill rates in seniors with hypertension. Am J Manag Care. 2009 Jan;15(1):59-66. PMID 19146365
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Babamoto KS, Sey KA, Camilleri AJ, Karlan VJ, Catalasan J, Morisky DE. Improving diabetes care and health measures among hispanics using community health workers: results from a randomized controlled trial. Health Educ Behav. 2009 Feb;36(1):113-26. doi: 10.1177/1090198108325911. PMID 19188371
- [Background] Cohen JL, Mann DM, Wisnivesky JP, Home R, Leventhal H, Musumeci-Szabo TJ, Halm EA. Assessing the validity of self-reported medication adherence among inner-city asthmatic adults: the Medication Adherence Report Scale for Asthma. Ann Allergy Asthma Immunol. 2009 Oct;103(4):325-31. doi: 10.1016/s1081-1206(10)60532-7. PMID 19852197
- [Background] Kripalani S, Risser J, Gatti ME, Jacobson TA. Development and evaluation of the Adherence to Refills and Medications Scale (ARMS) among low-literacy patients with chronic disease. Value Health. 2009 Jan-Feb;12(1):118-23. doi: 10.1111/j.1524-4733.2008.00400.x. PMID 19911444
- [Background] Hibbard JH, Mahoney E. Toward a theory of patient and consumer activation. Patient Educ Couns. 2010 Mar;78(3):377-81. doi: 10.1016/j.pec.2009.12.015. Epub 2010 Feb 25. PMID 20188505
- [Background] Hibbard JH, Mahoney ER, Stock R, Tusler M. Do increases in patient activation result in improved self-management behaviors? Health Serv Res. 2007 Aug;42(4):1443-63. doi: 10.1111/j.1475-6773.2006.00669.x. PMID 17610432
- [Background] Hibbard JH, Mahoney ER, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure. Health Serv Res. 2005 Dec;40(6 Pt 1):1918-30. doi: 10.1111/j.1475-6773.2005.00438.x. PMID 16336556
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Background] Anderson RM, Funnell MM, Fitzgerald JT, Marrero DG. The Diabetes Empowerment Scale: a measure of psychosocial self-efficacy. Diabetes Care. 2000 Jun;23(6):739-43. doi: 10.2337/diacare.23.6.739. PMID 10840988
- [Background] Anderson RM, Funnell MM, Nwankwo R, Gillard ML, Oh M, Fitzgerald JT. Evaluating a problem-based empowerment program for African Americans with diabetes: results of a randomized controlled trial. Ethn Dis. 2005 Autumn;15(4):671-8. PMID 16259492
- [Background] Tang TS, Funnell MM, Brown MB, Kurlander JE. Self-management support in "real-world" settings: an empowerment-based intervention. Patient Educ Couns. 2010 May;79(2):178-84. doi: 10.1016/j.pec.2009.09.029. Epub 2009 Nov 3. PMID 19889508
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Cleary PD, Jette AM. The validity of self-reported physician utilization measures. Med Care. 1984 Sep;22(9):796-803. doi: 10.1097/00005650-198409000-00003. PMID 6492908
- [Background] Ritter PL, Stewart AL, Kaymaz H, Sobel DS, Block DA, Lorig KR. Self-reports of health care utilization compared to provider records. J Clin Epidemiol. 2001 Feb;54(2):136-41. doi: 10.1016/s0895-4356(00)00261-4. PMID 11166528
- [Background] Reijneveld SA, Stronks K. The validity of self-reported use of health care across socioeconomic strata: a comparison of survey and registration data. Int J Epidemiol. 2001 Dec;30(6):1407-14. doi: 10.1093/ije/30.6.1407. PMID 11821355
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Baker DW, Williams MV, Parker RM, Gazmararian JA, Nurss J. Development of a brief test to measure functional health literacy. Patient Educ Couns. 1999 Sep;38(1):33-42. doi: 10.1016/s0738-3991(98)00116-5. PMID 14528569
- [Background] Davis TC, Michielutte R, Askov EN, Williams MV, Weiss BD. Practical assessment of adult literacy in health care. Health Educ Behav. 1998 Oct;25(5):613-24. doi: 10.1177/109019819802500508. PMID 9768381
- See also: Cellular Telecommunications and Internet Association. Semi-Annual Wireless Industry survey. Washington 2006. — https://www.ctia.org
- See also: Smith A. Mobile Access 2010. Pew Internet and American Life Project. 2010 — https://www.pewresearch.org/internet/2010/07/07/mobile-access-2010-2/
- See also: Fox S. Mobile Health 2010. Pew Internet and American Life Project. 2010 — https://www.pewinternet.org/wp-content/uploads/sites/9/media/Files/Reports/2010/PIP_Mobile_Health_2010.pdf